CLINICAL TRIAL: NCT07244211
Title: Musculoskeletal Adaptive Platform Trial (MAPT): Fixation Versus Arthroplasty Surgical Treatments for Early Recovery After HIP Fracture (FASTER-HIP)
Brief Title: MAPT Protocol: Fixation Versus Arthroplasty Surgical Treatments for Early Recovery After HIP Fracture (FASTER-HIP)
Acronym: FASTER-HIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); McMaster University (Other); University of Maryland, Baltimore (Other); Evellere Group (Unknown)
Responsible Party: Principal Investigator, Joseph Patterson, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPS-2024C1-37436; BPS-2024C1-37436 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2025-10-31; First posted 2025-11-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Femoral Neck Fractures
Keywords: Minimally displaced femoral neck fractures; arthroplasty; hip fractures; femoral fractures; orthopaedic procedures; older adults; patient-centered outcomes; adaptive trial; internal fixation; pragmatic trial
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures; Femoral Fractures | interventions — Arthroplasty, Replacement, Hip; Fracture Fixation, Internal

STUDY DESIGN:
Masking Description: The participant, treating clinicians, the research team, and the outcome assessors will not be blinded to the treatment allocation and outcome assessments. The data analysts and those interpreting the results of the trial will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip arthroplasty (Active Comparator)
  Interventions: Procedure: Hip arthroplasty
- Internal fixation (Active Comparator)
  Interventions: Procedure: Internal fixation

INTERVENTIONS:
Procedure: Hip arthroplasty — Participants will undergo surgical treatment using standard hip arthroplasty techniques for femoral minimally displaced femoral neck fracture. A modern porous-coated press-fit or cemented hip arthroplasty prosthesis will be used at the treating surgeon's discretion. Press-fit implants that have no ingrowth or ongrowth surface will not be permitted. The type of hip prosthesis (hemiarthroplasty or total hip arthroplasty), bearing (single or dual mobility), or the method of arthroplasty fixation (cemented or uncemented) will be at the discretion of the treating surgeon.
  Arms: Hip arthroplasty
Procedure: Internal fixation — Participants will undergo surgical treatment using standard fixation techniques for minimally displaced femoral neck fractures. The treating surgeon may perform fracture reduction maneuvers if desired. Fixed-angle devices and multiple screws will be permitted. The internal fixation device(s) will be inserted through a small lateral incision. Internal fixation constructs combining cancellous screws and fixed-angle devices will be permitted.
  Arms: Internal fixation

SUMMARY:
This study is an intervention domain of the Musculoskeletal Adaptive Platform Trial. The primary goal of this pragmatic, randomized, open-label, comparative effectiveness trial is to evaluate if arthroplasty is superior to internal fixation when used to treat minimally displaced femoral neck fractures in older adults ≥60 years old. We hypothesize that arthroplasty will reduce death, preserve ambulation, increase days alive and out of hospital, and improve health status compared to internal fixation within 4 months and 12 months from randomization.

DETAILED DESCRIPTION:
The Musculoskeletal Adaptive Platform Trial (MAPT) is an adaptive platform trial protocol that enables the simultaneous evaluation of multiple interventions (i.e., intervention domains) within a consistent infrastructure. Each intervention being evaluated in the MAPT will have an intervention domain protocol that describes additional eligibility criteria, interventions, secondary outcomes, and statistical stopping rules. The overarching objective of the MAPT trial platform is to incrementally decrease decisional uncertainty and identify treatments that will optimize patient outcomes. The platform focuses on the comparative effectiveness of available treatment options.

Adult patients aged 60 years or older with a low-energy minimally displaced femoral neck fracture treated with surgery are eligible for the FASTER-HIP intervention domain. Nearly half of all elderly hip fractures are femoral neck fractures, and approximately 20% are minimally displaced. Internal fixation has remained the treatment of choice for these injuries because these fractures can be fixed in situ, and the surgical implants can be inserted with little surgical dissection. Patients treated with internal fixation experience high complication rates, with the pooled risk of reoperation and mortality each above 14%. Preliminary data have suggested arthroplasty for minimally displaced fractures may lead to better patient outcomes, including improved ambulation, fewer reoperations, and a lower risk of death compared to internal fixation. While the preliminary data supporting the use of arthroplasty for minimally displaced fractures is promising, the necessary evidence to make this practice change remains lacking.

FASTER-HIP is a pragmatic, randomized, open-label, comparative effectiveness trial comparing hip arthroplasty versus internal fixation for minimally displaced femoral neck fractures. Randomization in this domain occurs in a 1:1 ratio (hip arthroplasty:internal fixation). The primary outcome is a composite of death within 120 days, ambulation status at 120 days, and days alive and out of hospital within 120 days of randomization. The primary outcome will be hierarchically assessed using the Win ratio. Secondary outcomes include the same composite at 365 days, individual components of the composite, health-related quality of life (EQ-5D-5L), and pain scores during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older undergoing surgery due to a minimally displaced femoral neck fracture
* The patient has a health condition affecting physical mobility.
* Complete fracture of the femoral neck (AO/OTA 31B) confirmed with anteroposterior and lateral hip radiographs, computed tomography, or magnetic resonance imaging.
* Minimally displaced fracture that could be, in the judgment of the attending surgeon, managed with either arthroplasty or in situ internal fixation without reduction.
* Low energy injury mechanism.
* Surgeons with expertise in internal fixation and total hip arthroplasty or hemiarthroplasty are available to perform surgery.

Exclusion Criteria:

* The patient is not clinically suitable for either compared treatment.
* Expected injury survival of less than 12 months.
* Terminal illness with expected survival of less than 12 months.
* Incarceration.
* Unable to obtain informed consent due to language barriers.
* Unable to obtain informed consent because the legally authorized representative was unavailable.
* Problems, in the judgment of the study personnel, with maintaining follow-up with the patient.
* Currently enrolled in a study or intervention domain that does not permit co-enrollment.
* Prior enrollment in the specific platform trial intervention domain.
* Patient or legally authorized representative did not provide informed consent (declined participation).
* Eligible patient or legally authorized representative was not approached within the screening window (missed participant).
* Other reasons to exclude the patient, as approved by the data coordinating center.
* Associated lower extremity injury that prevents post-operative weight-bearing.
* Retained hardware around the hip that precludes either study treatment.
* Infection around the hip (soft tissue or bone).
* Pathologic fracture with a lytic lesion in the femoral neck that precludes internal fixation.
* Injury did not occur within 21 days of screening.
* Patient is too ill, in the judgment of the attending surgeon, for internal fixation.
* Patient is too ill, in the judgment of the attending surgeon, for arthroplasty.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of death, ambulation status, and days alive and out of hospital. | 120 days after randomization
  Death consists of time to all-cause mortality.
  Ambulation will be evaluated using an ordinal ranking of independence.
  Days alive and out of hospital will be calculated by subtracting the sum of days meeting one of two criteria below:
  * Days not alive.
  * Any day on which the participant had an overnight stay in a hospital, inpatient rehabilitation, skilled nursing facility, nursing home, inpatient mental health care facility, or long-term care facility.

SECONDARY OUTCOMES:
Composite outcome of death, ambulation status, and days alive and out of hospital. | 365 days after randomization
  Death consists of time to all-cause mortality.
  Ambulation will be evaluated using an ordinal ranking of independence.
  Days alive and out of hospital will be calculated by subtracting the sum of days meeting one of two criteria below:
  * Days not alive.
  * Any day on which the participant had an overnight stay in a hospital, inpatient rehabilitation, skilled nursing facility, nursing home, inpatient mental health care facility, or long-term care facility.
Death | 120 days post-randomization
  Death consists of time to all-cause mortality.
Death | 12 months post-randomization
  Death consists of time to all-cause mortality.
Ambulation status | 120 days post-randomization
  Ambulation will be evaluated using an ordinal ranking of independence
Ambulation status | 12 months post-randomization
  Ambulation will be evaluated using an ordinal ranking of independence
Days alive and out of hospital | 120 days post-randomization
  Days alive and out of hospital will be calculated by subtracting the sum of days meeting one of two criteria below:
  * Days not alive.
  * Any day on which the participant had an overnight stay in a hospital, inpatient rehabilitation, skilled nursing facility, nursing home, inpatient mental health care facility, or long-term care facility.
Days alive and out of hospital | 12 months post-randomization
  Days alive and out of hospital will be calculated by subtracting the sum of days meeting one of two criteria below:
  * Days not alive.
  * Any day on which the participant had an overnight stay in a hospital, inpatient rehabilitation, skilled nursing facility, nursing home, inpatient mental health care facility, or long-term care facility.
Health-related quality of life | 120 days days post-randomization
  EQ-5D-5L - Range: 0 to 1, Higher scores indicates better self-perceived health
Health-related quality of life | 12 months post-randomization
  EQ-5D-5L - Range: 0 to 1, Higher scores indicates better self-perceived health
Numeric Pain Rating Scale | During hospitalization in the first seven postoperative days
  The highest level of pain recorded daily in the participant's medical record - Range: 0-10, higher score indicates higher level of pain

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T Patterson, MD, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - University of California, Irvine, Irvine, California
  - Los Angeles General Medical Center, Los Angeles, California
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Undecided